CLINICAL TRIAL: NCT06765798
Title: Effect of Adding Neural Mobilization to Mulligan Technique in Chronic Tennis Elbow
Brief Title: Adding Neural Mobilization to Mulligan Technique for Treatment of Patients With Chronic Tennis Elbow
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Safaa Radi Saber (Other)
Responsible Party: Sponsor-Investigator, Safaa Radi Saber, Master degree student .Basic Science . Physical therapy . Cairo university, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005457
Record Dates: First submitted 2024-12-27; First posted 2025-01-09 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2024-12

CONDITIONS: Tennis Elbow
Keywords: Tennis Elbow; Mulligan mobilization with movement; Neural Mobilization
MeSH Terms: conditions — Tennis Elbow | interventions — Movement; Congresses as Topic

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- group A (Experimental): Group A received neural mobilization for radial nerve, mulligan mobilization with movement and conventional therapy
  Interventions: Other: Group A : receive neural mobilization for radial nerve , mulligan mobilization with movement and conventional Therapy
- group B (Experimental): Group B received neural mobilization for radial nerve and conventional therapy
  Interventions: Other: Group B receive neural mobilization for radial nerve and conventional
- Group C (Experimental): Group C received mulligan mobilization with movement and conventional therapy
  Interventions: Other: Group C receive Mulligan mobilization with movement and conventional
- Group D (Active Comparator): Group D received conventional therapy
  Interventions: Other: Group D receive conventional

INTERVENTIONS:
Other: Group A : receive neural mobilization for radial nerve , mulligan mobilization with movement and conventional Therapy — Group A :Neural Mobilization for radial nerve, Mulligan Mobilization with Movement and Conventional neural mobilization for radial nerve: The physiotherapist holds the patient's arm and wrist while the patient reclined on his side then depress the shoulder, extend the elbow and then internally rotated the patient's arm. The patient's wrist, thumb, and fingers were all flexed, and the patient's ulnar was brought to deviation. While the patient's position was maintained, and the arm was abducted and then contralateral cervical side bending Mulligan mobilization with movement manual lateral glide MWM with gripping: Patient: Supine with upper limb fully supported on a treatment table. Treated body part: Relaxed extension of the elbow, shoulder internal rotation, with pronation of the forearm. Hands loosely around the grip dynamometer handles. Apply 6-10 repetitions in a set, with 3-5 sets in a treatment session, conventional ; Ultrasound therapy , stretching and strengthening for
  Arms: group A
Other: Group B receive neural mobilization for radial nerve and conventional — Group B receive neural mobilization for radial nerve and conventional neural mobilization for radial nerve: The physiotherapist holds the patient's arm and wrist while the patient reclined on his side then depress the shoulder, extend the elbow and then internally rotated the patient's arm. The patient's wrist, thumb, and fingers were all flexed, and the patient's ulnar was brought to deviation. While the patient's position was maintained, and the arm was abducted and then contralateral cervical side bending conventional ; Ultrasound therapy , stretching and strengthening for wrist flexors and extensors
  Arms: group B
Other: Group C receive Mulligan mobilization with movement and conventional — Group C receive Mulligan mobilization with movement and conventional
  Mulligan mobilization with movement manual lateral glide MWM with gripping: Patient: Supine with upper limb fully supported on a treatment table. Treated body part: Relaxed extension of the elbow, shoulder internal rotation, with pronation of the forearm. Hands loosely around the grip dynamometer handles. Apply 6-10 repetitions in a set, with 3-5 sets in a treatment session, conventional ; Ultrasound therapy , stretching and strengthening for wrist flexors and extensors
  Arms: Group C
Other: Group D receive conventional — Group D receive conventional :
  Ultrasound therapy , stretching and strengthening for wrist flexors and extensors
  Arms: Group D

SUMMARY:
The study aimed to assess the combined effect of neural mobilization and mulligan technique on pain ,functional disability and grip strength in patients with tennis elbow

DETAILED DESCRIPTION:
Tennis elbow, known as lateral epicondylitis (LE) describes an overuse injury secondary to an eccentric overload of the common extensor tendon at the origin of the extensor carpi radialis brevis (ECRB) tendon. Tennis elbow primarily results from the repetitive strain caused by activities that involve loaded and repeated gripping and/or wrist extension. It is common in individuals who play tennis, squash, badminton, or any activity involving repetitive wrist extension, radial deviation, and/or forearm supination.

Patients with tennis elbow usually report pain or tenderness at the lateral epicondyle of the humerus, decreased gripping strength, and weakness when turning their palms up and straightening their wrists. Pain and inflammation of make it difficult to move the elbow joint through its full range of motion because of the pain and affect function of joint (ECRB)

Radial nerve mobilization exercises, has been used to treat musculoskeletal problems, including LE. Nerve mobilization or neurodynamic mobilization, defined by David Butler, is aimed at restoring homeostasis in and around the nervous system through facilitating movement between neural structures and their surroundings. It is stated that neural shifting reduces adhesions between the nerve and surrounding tissue, improves neural vascularity, and improves the axoplasmic flow Mulligan mobilization with movement (MWM) is a form of manual therapy that includes a sustained lateral glide to the elbow joint with concurrent physiological movement. This mobilization technique is often used to correct the faulty position of the elbow joint. It is the primary modality for the correction of positional fault of the elbow joint complex mimicking a contractile element pathology of the common extensor bundle." Which result in reducing pain, improvement of pain-free grip strength (PFGS), and increased ability to tolerate resisted isometric wrist extension

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 20-60 years old

  * . Diagnosed with chronic tennis elbow
  * experienced discomfort in their dominant arm, tenderness over the lateral epicondyle of the elbow joint, and exhibited signs and symptoms of tennis elbow persisting for three months
  * Increased pain with resistant elbow extension, wrist extension, gripping, and supination
  * ULTT 2 b (radial nerve) should be positive ) pain referral throughout the dorsal and radial aspect of the forearm and, sometimes, an "electrical shock-like" pain on the radial side of the right wrist (

Exclusion Criteria:

* patients who had a history of or were suffering from psychogenic stress

  * acute strain, fractures of the humerus, radius, and ulna,
  * History of Rheumatoid diseases
  * Subjects on steroids or any other medications for pain at present were excluded
  * severe edema, infection
  * malignancy
  * osteoporosis
  * unstable joints
  * severe neck or shoulder pain, neurological conditions \ impacting the upper extremity Cervical radiculopathy
  * Bilateral Symptoms of Tennis elbow

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
pain by visual analgue scale | from enrollment to the end of treatment at 4 weeks , assessment will be done pre and post treatment
  pain will be assessed by visual analogue scale (VAS) which involves having them mark along a 10 cm-long line with a number ranging from 0 to 10. "0" denotes no discomfort, and "10" denotes the most agonizing pain possible They are generally completed by patients themselves. The patients marks on the line the point that they feel represents their perception of their current state of pain.
Functional disability | from enrollment to the end of treatment at 4 weeks , assessment will be done pre and post treatment
  Functional Disability will be assessed by Arabic version of DASH Questionnaire DASH Arabic contains 30 items, like the original DASH, each item has five response choices that range from 1, ''without any difficulty or no symptoms exist'' to 5, ''unable to engage in activity or very severe symptoms''. In order for a score to be calculated, a minimum of 27 of the 30 items must be completed. The assigned values for all completed responses are added and averaged to yield a score of 5 or less; this value is then transformed to 100 by subtracting 1 and multiplying by 25, to make it easy to compare with other measures that are scaled from 0 to 100: the higher the score, the greater the disability
Maximum grip strength | from enrollment to the end of treatment at 4 weeks , assessment will be done pre and post treatment
  Maximum grip strength by Jamer hand dynamometer The gold standard for measuring grip strength is the JAMAR® Hydraulic Hand Dynamometer. Where possible, participants were positioned sitting upright in a chair, with their knees and hips at 90° and with back support. For those unable to mobilize out of bed, the head of the bed was raised as far as possible, ensuring an upright long-sitting position. The shoulder on the dominant side was adducted against the body, the elbow positioned in 90° flexion (unsupported) and the wrist in a neutral position. Participants were then instructed to grip the dynamometer as strongly as they possibly could, using their dominant hand .The measurements of both extremities were repeated 3 times with resting interval of 30 s between each measurement. The average of the three trials was recorded in kilograms (kg).

CONTACTS AND LOCATIONS:
Overall Officials: Maher Ahmed Elkeblawy Professor of physical Therapy,Department of Basic Science, Professor of physical Therapy, Study Director — Professor of physical Therapy ,Department of Basic Science , Faculty of Physical Therapy Cairo University; Mariam Omran Grace Lecturer of Physical Therapy .Basic Science . cairo university, Lecturer of Physical Therapy ., Study Director — Lecturer of Physical Therapy .Basic Science . cairo university; Mohamed Ali Hashish Lecturer of orthopedic and spine surgery, Cairo university,, Lecturer, Study Director — Lecturer of orthopedic and spine surgery , Cairo university ,kasr Al-ainy
Locations (1):
- Delta University, Gamasa, Egypt

IPD SHARING:
Plan to Share IPD: No